CLINICAL TRIAL: NCT01828827
Title: A Phase 1, Randomized, Balanced, Single-Dose, Two-Treatment, Two-Period, Two-Sequence, Crossover, Open-Label Study of the Effect of Food on the Bioavailability and Pharmacokinetics of PA-824 Tablets in Healthy Adult Subjects
Brief Title: Food Effect Study on the Bioavailability and PK of PA-824 Tablets in Healthy Adult Subjects
Acronym: CL-003
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: PA-824 CL-003
Record Dates: First submitted 2013-02-12; First posted 2013-04-11 (Estimated); Last update posted 2016-01-14 (Estimated); Status verified 2015-08

CONDITIONS: Tuberculosis
Keywords: tuberculosis; PK; PA-824; food effect,; bioavailability; pretomanid; CL-003
MeSH Terms: conditions — Tuberculosis | interventions — pretomanid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fed 1000 mg PA-824 (Experimental): Each dose will be 1000 mg PA-824 (5 x 200 mg tablets), and will be administered with 240 mL tap water approximately 30 minutes after a high-calorie, high-fat breakfast provided after a minimum 10-hour overnight fast.
  Interventions: Drug: PA-824 1000 mg
- Fasting 1000 mg PA-824 (Experimental): Each dose will be 1000 mg PA-824 (5 x 200 mg tablets), and will be administered with 240 mL tap water after a minimum 10-hour overnight fast.
  Interventions: Drug: PA-824 1000 mg

INTERVENTIONS:
Drug: PA-824 1000 mg — Two single administrations of 1000mg each administered by 5 tablets of 200mg, one administered in the fed state and one administered in the fasted state.

SUMMARY:
This is a Phase 1, single-center, randomized, balanced, single-dose, two-treatment, two-period, two-sequence, crossover, open-label study to evaluate the effect of food on the pharmacokinetics of PA-824. This study was designed to understand the possible effects of a high-calorie, high-fat meal on PA-824 absorption and pharmacokinetics. The hypothesis to be tested in this study is that the rate and extent of absorption of PA-824, as measured by Tmax, Cmax, AUC(0-t), and AUC(0 inf), are the same after a high-calorie, high-fat meal as compared with after a minimum 10-hour fast.

ELIGIBILITY:
Inclusion Criteria:

1. Have the ability to understand the requirements of the study, have provided written informed consent (as evidenced by signature on an informed consent document approved by an IRB), and agree to abide by the study restrictions.
2. Be healthy non-tobacco/nicotine using (6-month minimum) adult subjects, 19 to 50 years of age, inclusive.
3. Be medically healthy subjects with clinically insignificant Screening results (among laboratory profiles, medical histories, ECGs, or physical exam), as deemed by the Principal Investigator.
4. Have a body mass index of 18 to 29.
5. Have negative urine test results for alcohol and drugs of abuse such as amphetamines, cannabinoids, and cocaine metabolites at both Screening and Check-in.
6. Agree to follow the requirements set forth in the protocol regarding pregnancy controls and donation of sperm, blood, or blood components.

Exclusion Criteria:

1. Any clinically significant (as deemed by the Principal Investigator) history, acute illness (resolved within 4 weeks of screening), or presence of cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal (including eating disorders), endocrine, metabolic, immunologic, dermatologic, neurologic, psychological, or psychiatric disease.
2. Any serum creatinine or BUN measure beyond the upper limit of the normal range at Screening or Check-in. Individual values may be discussed with the Sponsor Medical Monitor.
3. Positive Screening test for HCV, HBV, or HIV.
4. History of peptic ulcer disease, gastritis, esophagitis, or gastroesophageal reflux disease.
5. History of any cardiac abnormality (as deemed by the Principal Investigator).
6. History of hypokalemia or hypomagnesemia.
7. History of prolonged QT interval.
8. Family history of Long-QT Syndrome or sudden death without a preceding diagnosis of a condition that could be causative of sudden death (such as known coronary artery disease or CHF or terminal cancer)
9. Resting pulse rate < 40 or > 100 bpm at Screening.
10. At either Screening or the pre-dose read before the first dose, a QTcB (Bazett's correction) >430 msec, calculated from the average of triplicate reads collected at one sitting.
11. At either Screening or the pre-dose read before the first dose, a QTcF (Fridericia's correction) >430 msec, calculated from the average of triplicate reads collected at one sitting.
12. History or presence of alcoholism or drug abuse within the past 2 years (as deemed by the Principal Investigator).
13. Use of alcohol within 72 hours prior to dosing.
14. Significant history of drug and/or food allergies (as deemed by the Principal Investigator).
15. For women, lactation.
16. For women, positive test for serum HCG at Screening or Check-in.
17. Use of any systemic or topical prescription medication within 14 days prior to dosing or during the study, except hormonal contraceptives in women.
18. Use of any systemic or over-the-counter medication including vitamins, herbal preparations, antacids, cough and cold remedies, etc., within 7 days prior to dosing or during the study.
19. Use of any drugs or substances within 30 days prior to dosing known to be strong inhibitors or inducers of cytochrome P450 enzymes (including xenobiotics, quinidine, tyramine, ketoconazole, testosterone, quinine, gestodene, metyrapone, phenelzine, doxorubicin, troleandomycin, cyclobenzaprine, erythromycin, cocaine, furafylline, cimetidine, dextromethorphan, etc.) or known to prolong the QT interval (including amiodarone, bepridil chloroquine, chlorpromazine, cisapride, clarithromycin, disopyramide dofetilide, domperidone, droperidol, erythromycin, halofantrine, haloperidol, ibutilide, levomethadyl, mesoridazine, methadone, pentamidine, pimozide, procainamide, quinidine, sotalol, sparfloxacin, thioridazine, etc.).
20. Use of any therapeutic agents known to alter any major organ function (e.g., barbiturates, opiates, phenothiazines, cimetidine, etc.) within 30 days prior to dosing.
21. Consumption of products containing grapefruit within 10 days prior to dosing.
22. Any special dietary changes during the 30 days prior to dosing, as deemed by the Principal Investigator in consultation with the Sponsor Medical Monitor.
23. Any strenuous exercise within 7 days of Check-in, as deemed by the Principal Investigator in consultation with the Sponsor Medical Monitor.
24. Donation of whole blood or significant loss of blood within 56 days prior to dosing.
25. Plasma donation within 7 days prior to dosing.
26. Participation in another interventional clinical trial within 30 days prior to dosing.
27. Hemoglobin < 12.0 g/dL.
28. Previous use of PA-824.
29. Any other factor which suggests to the Principal Investigator that the subject should not participate in the study.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2007-03; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Time of maximum drug concentration in hours [Tmax] | mean through 168 hours after each dose with measurements at predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, 24, 30, 36, 48, 72, 96, 120, 144 and 168 hours post dose
  To compare the rate and extent of absorption as measured by Tmax of a single 1000 mg oral dose of PA-824 tablets in healthy adult male and female subjects when PA-824 is administered after a high-calorie, high-fat meal and when it is administered after a minimum 10-hour fast. Tmax is obtained without interpolation.
Maximum observed drug concentration in ng/mL [Cmax] | mean through 168 hours after each dose with measurements at predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, 24, 30, 36, 48, 72, 96, 120, 144 and 168 hours post dose
  To compare the rate and extent of absorption as measured by Cmax of a single 1000 mg oral dose of PA-824 tablets in healthy adult male and female subjects when PA-824 is administered after a high-calorie, high-fat meal and when it is administered after a minimum 10-hour fast.
Area under the drug concentration-time curve in ng*hour/mL [AUC0-t] | mean through 168 hours after each dose with measurements at predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, 24, 30, 36, 48, 72, 96, 120, 144 and 168 hours post dose
  To compare the rate and extent of absorption as measured by AUC0-t of a single 1000 mg oral dose of PA-824 tablets in healthy adult male and female subjects when PA-824 is administered after a high-calorie, high-fat meal and when it is administered after a minimum 10-hour fast. AUC(0-t) is calculated using linear trapezoidal summation from time zero to time t, where t is the time of the last measurable concentration.
Area under the drug concentration-time curve from time zero to infinity in ng*hour/mL [AUC(0-inf)] | mean through 168 hours after each dose with measurements at predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, 24, 30, 36, 48, 72, 96, 120, 144 and 168 hours post dose
  To compare the rate and extent of absorption as measured by AUC0-inf of a single 1000 mg oral dose of PA-824 tablets in healthy adult male and female subjects when PA-824 is administered after a high-calorie, high-fat meal and when it is administered after a minimum 10-hour fast. AUC(0-inf) is calculated as AUC(0-t) + Ct/Kel.

SECONDARY OUTCOMES:
Ratio of AUC(0-t) to AUC(0-inf) [AUC(0-t)/ AUC(0-inf)] | mean through 168 hours after each dose with measurements at predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, 24, 30, 36, 48, 72, 96, 120, 144 and 168 hours post dose
  To compare additional pharmacokinetic (PK) parameters such as AUC(0-t)/ AUC(0-inf) of a single 1000 mg oral dose of PA-824 tablets in healthy adult male and female subjects when PA-824 is administered after a high-calorie, high-fat meal and when it is administered after a minimum 10-hour fast.
Number of participants with adverse events | through the study (Day 1-Day 17)
  To compare the safety and tolerability as measured by the number of participants with adverse events after a single 1000-mg oral dose of PA-824 tablets in healthy adult male and female subjects when PA-824 is administered after a high-calorie, high-fat meal and when it is administered after a minimum 10-hour fast.
Elimination half-life in hours [t1/2] | mean through 168 hours after each dose with measurements at predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, 24, 30, 36, 48, 72, 96, 120, 144 and 168 hours post dose
  To compare additional pharmacokinetic (PK) parameters such as t1/2 of a single 1000 mg oral dose of PA-824 tablets in healthy adult male and female subjects when PA-824 is administered after a high-calorie, high-fat meal and when it is administered after a minimum 10-hour fast. T1/2 is calculated as ln (2)/Kel.
Terminal elimination rate constant in 1/hour [Kel] | mean through 168 hours after each dose with measurements at predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, 24, 30, 36, 48, 72, 96, 120, 144 and 168 hours post dose
  To compare additional pharmacokinetic (PK) parameters such as Kel of a single 1000 mg oral dose of PA-824 tablets in healthy adult male and female subjects when PA-824 is administered after a high-calorie, high-fat meal and when it is administered after a minimum 10-hour fast. Kel is calculated by linear regression of the terminal linear portion of the log concentration vs. time curve.
Oral clearance in L/hour (Cl/F) | mean through 168 hours after each dose with measurements at predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, 24, 30, 36, 48, 72, 96, 120, 144 and 168 hours post dose
  To compare additional pharmacokinetic (PK) parameters such as Cl/F of a single 1000 mg oral dose of PA-824 tablets in healthy adult male and female subjects when PA-824 is administered after a high-calorie, high-fat meal and when it is administered after a minimum 10-hour fast. Cl/F is calculated as dose/AUC(0-inf).
Volume of distribution in L (Vd/F) | mean through 168 hours after each dose with measurements at predose, 0.5, 1, 2, 3, 4, 5, 6, 7, 8, 12, 16, 24, 30, 36, 48, 72, 96, 120, 144 and 168 hours post dose
  To compare additional pharmacokinetic (PK) parameters such as Vd/F of a single 1000 mg oral dose of PA-824 tablets in healthy adult male and female subjects when PA-824 is administered after a high-calorie, high-fat meal and when it is administered after a minimum 10-hour fast. Vd/F is calculated as the ratio of CL/F/Kel.

CONTACTS AND LOCATIONS:
Overall Officials: C James Kissling, MD, Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Lincoln, Nebraska, United States

REFERENCES:
- [Derived] Winter H, Ginsberg A, Egizi E, Erondu N, Whitney K, Pauli E, Everitt D. Effect of a high-calorie, high-fat meal on the bioavailability and pharmacokinetics of PA-824 in healthy adult subjects. Antimicrob Agents Chemother. 2013 Nov;57(11):5516-20. doi: 10.1128/AAC.00798-13. Epub 2013 Aug 26. PMID 23979737
- See also: Global Alliance for TB Drug Development website — http://www.tballiance.org